CLINICAL TRIAL: NCT07177105
Title: Primary Tumor Resection Combined With Sintilimab and Chemotherapy for Advanced Non-small-cell Lung Cancer: A Randomized Controlled Trial
Brief Title: Primary Tumor Resection With Sintilimab and Chemotherapy in Advanced NSCLC
Acronym: SURGAN-ICI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jianxing He (Other)
Responsible Party: Sponsor-Investigator, Jianxing He, The First Affiliated Hospital of Guangzhou Medical University, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-2025-159-02
Record Dates: First submitted 2025-09-06; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Sintilimab; Chemotherapy; Surgery; Advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Active Comparator): Participants will first undergo cytoreductive surgery. After adequate postoperative recovery within 2-4 weeks, they will receive therapy consisting of intravenous administration of sintilimab, pemetrexed, and carboplatin on Day 1 of each 3-week cycle, for a total of 4 cycles. During the maintenance phase, participants will receive sintilimab and pemetrexed until the duration of sintilimab treatment reaches 31 cycles, or the total treatment duration from randomization reaches 2 years, or until disease progression or the occurrence of unacceptable toxicity.
  Interventions: Drug: Immunochemotherapy
- Intervention Group (Experimental): Participants will receive induction therapy consisting of intravenous administration of sintilimab, pemetrexed, and carboplatin on Day 1 of each 3-week cycle, for a total of 4 cycles. During the maintenance phase, participants will receive sintilimab and pemetrexed until the duration of sintilimab treatment reaches 31 cycles, or the total treatment duration from randomization reaches 2 years, or until disease progression or the occurrence of unacceptable toxicity.
  Interventions: Procedure: Cytoreductive surgery; Drug: Immunochemotherapy

INTERVENTIONS:
Procedure: Cytoreductive surgery — * Preoperative evaluation must confirm resectability. Thoracoscopic minimally invasive surgery will be performed, with the surgical approach selected according to disease conditions, such as lobectomy, segmentectomy, wedge resection, or sleeve resection; ② Systematic mediastinal lymph node dissection or lymph node sampling (based on preoperative imaging and intraoperative evaluation) must be performed; ③ Postoperative recovery must be adequate (postoperative complications ≤ Clavien-Dindo grade II).
  Arms: Intervention Group
Drug: Immunochemotherapy — 1. Treatment phase:
     ① Sintilimab Dose: 200 mg, administered intravenously over 30 minutes or less;
     ② Pemetrexed Dose: 500 mg/m², administered intravenously over 10 minutes or less;
     ③ Carboplatin Dose: administered according to the area under the curve (AUC) of 5 mg/mL/min, with infusion time controlled within 15-60 minutes.
     The above regimen will be administered every 3 weeks after surgery for a total of 4 cycles.
  2. Maintenance phase:
     * Sintilimab Dose: 200 mg, administered intravenously over 30 minutes or less; ② Pemetrexed Dose: 500 mg/m², administered intravenously over 10 minutes or less; The above regimen will be administered every 3 weeks. Maintenance with sintilimab will continue for up to 31 cycles, or the total duration of systemic therapy from randomization will not exceed 2 years, or until disease progression or the occurrence of unacceptable toxicity

SUMMARY:
This study aims to evaluate whether resecting the primary tumor can improve the outcomes of treatment with sintilimab and chemotherapy in advanced EGFR/ALK-negative non-small cell lung cancer (NSCLC). Patients will be randomly assigned to one of two groups: one group will undergo primary tumor resection followed by sintilimab, pemetrexed, and carboplatin, while the other group will only receive sintilimab, pemetrexed, and carboplatin. The study will assess progression-free survival, overall survival, treatment response, safety, and the impact of treatment on quality of life. Through this study, we hope to determine whether primary tumor resection can provide additional benefits of anti-PD-1 therapy and chemotherapy for advanced NSCLC.

DETAILED DESCRIPTION:
This study is a single-center, randomized, open-label, parallel-group trial designed to evaluate the efficacy and safety of primary tumor resection combined with sintilimab, pemetrexed, and carboplatin in patients with advanced, EGFR/ALK-negative NSCLC. A total of 118 patients will be enrolled and randomly assigned in a 1:1 ratio to one of two treatment groups: one group will receive tumor resection followed by the combination of sintilimab, pemetrexed, and carboplatin, while the other group will receive sintilimab, pemetrexed, and carboplatin without tumor resection. The primary endpoint of the study is progression-free survival (PFS), as assessed by independent radiological review according to RECIST v1.1 criteria. Secondary outcomes include overall survival (OS), objective response rate (ORR), disease control rate (DCR), adverse effects (AEs), serious adverse effects (SAEs) and quality of life (QoL). Statistical analysis will include Kaplan-Meier estimation of median PFS with 95% confidence intervals, log-rank testing for comparing differences between the two treatment groups, and Cox proportional hazards models for calculating hazard ratios. Stratification will be performed based on clinical stage, histological subtype, PD-L1 expression, tumor size, and baseline demographic characteristics. Patients will be followed up until disease progression or death from randomization. The results of this study will provide valuable insights into the potential benefits of combining surgery with anti-PD-1 therapy and chemotherapy for advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, no sex limitation;
2. Histologically or cytologically confirmed stage III-IV non-squamous NSCLC, deemed unresectable (evaluated by MDT);
3. Negative for EGFR mutation and ALK rearrangement (tested by ARMS-PCR, NGS, or equivalent methods);
4. No histological evidence of small cell lung cancer (SCLC) or transformation to SCLC;
5. No prior exposure to anti-tumor therapy;
6. ECOG performance status of 0-1;
7. Expected survival ≥ 6 months;
8. Primary tumor diameter ≥ 1 cm, with at least one measurable lesion remaining after resection (per RECIST v1.1 criteria);
9. Adequate major organ function, including:

   ① Hematologic: absolute neutrophil count ≥ 1.5 × 10⁹/L, platelets ≥ 100 × 10⁹/L, hemoglobin ≥ 9.0 g/dL;

   ② Hepatic: ALT and AST ≤ 2.5 × ULN (≤ 5 × ULN in case of liver metastases), total bilirubin ≤ 1.5 × ULN;
   * Renal: serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min (calculated by Cockcroft-Gault formula);
10. Pulmonary function (patients must meet at least one of the following to ensure adequate postoperative pulmonary reserve):

    ① FEV1 ≥ 1.2 L (or ≥ 40% of predicted value);

    ② FEV1/FVC ≥ 0.7, excluding severe obstructive ventilatory impairment;

    ③ DLCO (diffusing capacity for carbon monoxide) ≥ 40% of predicted value, to assess diffusion capacity;

    ④ If preoperative FEV1 < 1.2 L or DLCO < 40%, a quantitative perfusion scan is recommended along with preoperative exercise testing (e.g., 6-minute walk test, stair-climbing test) to evaluate residual pulmonary function;
11. Preoperative assessment by the study team confirming that the patient can tolerate primary lesion resection;
12. Signed informed consent with willingness to comply with study protocol.

Exclusion Criteria:

1. Impaired immune function: history of primary immunodeficiency; history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
2. Active brain metastases. Patients with adequately treated brain metastases may be eligible if they have remained neurologically stable for at least 2 weeks prior to study entry and are not receiving systemic corticosteroids or are on a stable/reducing dose equivalent to ≤10 mg prednisone daily.
3. Pregnancy.
4. Presence of any severe, uncontrolled, or unstable comorbidity that, in the opinion of the investigator, may interfere with the patient's participation in the study or affect the interpretation of study results, including uncontrolled seizures, psychiatric disorders, active or uncontrolled infections, or other conditions (including laboratory abnormalities).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization until the first documentation of disease progression or death from any cause, whichever occurs first (up to 5 years).
  PFS is defined as the time from randomization to the first documentation of disease progression (PD) or death from any cause, whichever occurs first. Disease progression will be assessed by the Independent Radiology Review Committee (IRRC) according to RECIST version 1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | Randomization to death from any cause (up to 5 years).
  OS is defined as the time from randomization to death from any cause.
Objective Response Rate (ORR) | Randomization until disease progression or death, which ever occurs first (up to 5 years).
  The proportion of patients achieving complete and partial remission after treatment, measured according to RECIST v1.1 criteria.
Disease Control Rate (DCR) | Randomization until disease progression or death, which ever occurs first (up to 5 years).
  DCR is defined as the proportion of participants with complete response, partial response, and stable disease, as determined by RECIST v1.1 criteria.
Adverse Events | Randomization up to approximately 5 years.
  Safety will be assessed by recording treatment-related adverse events (AEs) and serious adverse events (SAEs), graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Quality of Life (QoL) evaluated by European Organisation for Research and Treatment of Cancer core quality of life questionnaire (EORTC QLQ-C30) | Randomization until disease progression or death, which ever occurs first (up to 5 years).
  The EORTC QLQ-C30 is a 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients (range: 0-100; higher scores indicate better functioning and quality of life).
Quality of Life (QoL) evaluated by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module (EORTC QLQ-LC13) | Randomization until disease progression or death, which ever occurs first (up to 5 years).
  Supplementary lung cancer-specific questionnaire to be used in conjunction with the QLQ-C30 (range: 0-100; higher scores indicate worse lung cancer-related symptoms).

IPD SHARING:
Plan to Share IPD: No